## The Effect of the Check List Developed for Drug Administration From Enteral Nutrition Tube on Administration Errors

01.10.2022

The study was carried out on 69 subjects. The data was completed by transferring to IBM SPSS Statistics 23 program. While evaluating the study data, firstly the Kolmogorow-Smirnov test was applied for the normal distribution and it was decided to apply parametric tests. Descriptive statistics (mean, standard deviation) are given for numerical variables. Independent sample t-test and chi-square test were used for the difference between the two groups, and the dependent sample t-test was used to examine the differences between the times. P<0.05 was accepted for significance.